CLINICAL TRIAL: NCT00866983
Title: A Local, Multi-Centre, Extension, Open Label Access Study, To Provide Sildenafil Therapy For Patients Who Completed A1481244 Study And Are Judged By The Investigator To Derive Clinical Benefit From Continued Treatment With Sildenafil , Prior To Reimbursement And Availability For Patients In Brazil.
Brief Title: Local Open-Label Access Study For Patients Who Completed A1481244 Study In Brazil
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481270
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Open label; sildenafil; PAH; Brazil
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: sildenafil (Revatio) 20 mg TID — To provide access to sildenafil for patients completing the A1481244 study, resides in Brazilian States where Revatio™ is not supplied by Health Secretary and are judged by the Investigator to derive clinical benefit from continued treatment with sildenafil. It will be supplied until the patient gets access to Sildenafil through Brazilian State Health Secretary from where the patient resides.
  Other Names: sildenafil, Revatio

SUMMARY:
The purpose of this study is to provide sildenafil therapy to patients who completed the A1481244 study for the treatment of PAH, and reside in Brazilian States where Revatio™ is not supplied by Health Secretary, and are judged by the Investigator to derive clinical benefit from continued treatment with Sildenafil. It will be supplied until patient gets access to Sildenafil through Brazilian State Health Secretary from where patient resides.

ELIGIBILITY:
Inclusion Criteria:

* Subject who completed the A1481244 study and are judged by the Investigator to derive clinical benefit from continuous treatment with Sildenafil 20 mg therapy.
* Subject who resides in a Brazilian State where Sildenafil is not supplied by State Health Secretary.

Exclusion Criteria:

* Pregnant or lactating women.
* Current participation in other studies and during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Brazil (2):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481270&StudyName=Local%20Open-Label%20Access%20Study%20For%20Patients%20Who%20Completed%20A1481244%20Study%20In%20Brazil